CLINICAL TRIAL: NCT01605552
Title: Computer-Based Depression Treatment to Reduce Coronary Artery Disease Risk
Brief Title: Beating the Blues for Your Heart
Acronym: BtB-Heart
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Jesse Stewart, Assistant Professor of Psychology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1105005448; CRP4880000 (Other Grant/Funding Number: American Heart Association); 1703 (Other: Indiana Clinical Research Center)
Record Dates: First submitted 2012-05-09; First posted 2012-05-25 (Estimated); Results first posted 2016-02-24 (Estimated); Last update posted 2022-12-29 (Actual); Status verified 2022-11

CONDITIONS: Depression; Depressive Symptoms; Cardiovascular Disease (CVD); Coronary Artery Disease (CAD); Heart Disease
Keywords: Depression; Depressive Symptoms; Cardiovascular Disease (CVD); Coronary Artery Disease (CAD); Heart Disease
MeSH Terms: conditions — Depression; Cardiovascular Diseases; Coronary Artery Disease; Heart Diseases | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Beating the Blues (BtB) (Experimental): An 8-session, empirically supported, computerized, cognitive-behavioral intervention for depression (www.beatingthebluesus.com)
  Interventions: Behavioral: Beating the Blues (BtB)
- Usual Care (Other): Patients and their primary care providers were informed of the positive depression screen, and follow-up was encouraged.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Beating the Blues (BtB) — BtB is a widely used, empirically supported, computer-based, CBT program for depression designed for use in primary care clinics. BtB utilizes an interactive, multimedia format to deliver and eight 50-minute, weekly therapy sessions. General topics covered include identifying and challenging automatic thoughts, cognitive errors, core beliefs, and attributional styles; activity scheduling; problem solving; graded exposure; task breakdown; sleep management; and relapse prevention. In addition to session work, patients are assigned homeworks that are customized to their needs and reviewed at the start of each session. A progress report, including whether the patient is experiencing suicidal ideation, is generated at the end of each session.
  Other Names: Computer-Based Cognitive Behavioral Therapy (CBT); Computer-Based Psychotherapy
  Arms: Beating the Blues (BtB)
Other: Usual Care — Patients randomized to usual care will be informed that they have clinically significant depressive symptoms and will be encouraged to follow-up with their primary care physicians, who will receive a letter from our team indicating that their patient has elevated depressive symptoms and was randomized to the control condition. The letter will also encourage physicians to follow-up with their patients and will provide a list of local mental health services. Like those in the intervention group, usual care patients will continue to have access to and will receive any medical and mental health services that are part of usual care in the targeted health care systems. Thus, there are no restrictions regarding the care that these patients can receive.
  Other Names: Treatment As Usual (TAU)
  Arms: Usual Care

SUMMARY:
The objective of this clinical trial is to evaluate whether a computerized depression treatment, delivered before the onset of heart disease, reduces the risk of heart disease in the future. Participants in this trial will be primary care patients who are depressed but do not have a history of heart disease. Half of these patients will receive a standard treatment (usual care), and the other half will receive eight weeks of an evidence-based psychological treatment called Beating the Blues®, which is a computerized, cognitive behavioral treatment program for depression. To evaluate change in heart disease risk, the investigators will measure the functioning of the arteries using ultrasound before and after the treatment. It is hypothesized that patients who receive Beating the Blues® will show greater improvements in both depression and artery function than patients who receive standard treatment.

DETAILED DESCRIPTION:
Depression is an independent risk factor for coronary artery disease (CAD); unfortunately, past trials have not detected a cardiovascular benefit. A promising and unexplored explanation for these results is that the interventions were delivered too late in the natural history of CAD. Because no study has evaluated this possibility, there is a critical need to determine whether evidence-based depression treatment, delivered before the onset of clinical CAD, reduces cardiovascular risk. Accordingly, the objective of the proposed clinical and translational research is to perform a preliminary evaluation of the efficacy of a highly disseminable depression intervention in decreasing CAD risk. To achieve this goal, a clinical trial of depressed primary care patients free of cardiovascular disease is being conducted. Patients will be randomized to usual care or a computer-based, cognitive behavioral intervention called Beating the Blues®, the most widely used and empirically supported computerized treatment program for depression. The primary outcome is brachial artery flow-mediated dilation, a noninvasive measure of endothelial function. The specific aim of the proposed trial is to evaluate whether Beating the Blues®, delivered prior to the onset of clinical CAD, improves endothelial dysfunction. Demonstrating that earlier treatment of depression with Beating the Blues lowers CAD risk, the long-term expected outcome, would place computed-based depression treatment in the armamentarium of CAD prevention strategies of the primary care provider. This change to clinical practice should result in improved cardiovascular risk management, which in turn would translate into reduced CAD morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Primary care patients
* Age ≥40 years
* Clinically significant depressive symptoms (Patient Health Questionnaire-9 ≥10)
* No history of cardiovascular disease

Exclusion Criteria:

* Pregnant women
* A history of chronic disorders (HIV/AIDS, chronic kidney disease, systemic inflammatory disease, or past-year cancer)
* Current use of anticoagulants or vasodilators (antihypertensive and lipid-lowering medications are allowed)
* Current drinking problem
* History of bipolar disorder or psychosis
* Ongoing treatment for depression with a psychiatrist or psychologist/ counselor (antidepressants alone are allowed)
* Severe cognitive impairment
* Acute risk of suicide
* Significant vision or hearing problems
* Individuals who do not read or speak English

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesse C. Stewart, Ph.D., Principal Investigator — Indiana University-Purdue Univerisity Indianapolis
Locations (1):
- Indiana University-Purdue University Indianapolis (IUPUI), Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Beating the Blues (BtB) | Usual Care
Started | 13 | 16
Completed | 7 (4 dropped out before the first BtB visit; it is unlikely that the treatment was the cause of dropout) | 14
Not Completed | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Beating the Blues (BtB) | Usual Care | Total
Number analyzed (Participants) | 13 | 16 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (6.3) | 50.5 (6.7) | 49.2 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Post-Treatment Brachial Flow-Mediated Dilation (FMD) Adjusted for Pre-Treatment FMD
Description: Patients will undergo ultrasound assessment of brachial FMD in accordance with established guidelines. After a 10-minute supine rest, high-resolution baseline images of the brachial artery will be obtained from 3 consecutive cardiac cycles. Next, the forearm cuff will be inflated to 250 mmHg for 5 minutes and then will be rapidly deflated. At 60 and 90 seconds post-deflation, images from 3 consecutive cardiac cycles will be acquired. FMD values will be computed as the % change in brachial diameter at either 60 or 90 seconds after cuff deflation.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: % change in brachial diameter
Arm/Group | Beating the Blues (BtB) | Usual Care
Number analyzed (Participants) | 7 | 14
% change in brachial diameter | 4.18 (2.86) | 2.47 (2.72)
Statistical Analysis 1: Comparison: Beating the Blues (BtB) vs Usual Care; Test type: Superiority; p = .21, ANCOVA; Cohen's d = 0.61

2. Secondary Outcome: Post-Treatment Depressive Symptoms Severity (SCL-20 Score) Adjusted for Pre-Treatment SCL-20 Score
Description: Self-reported depressive symptom severity was measured at pre- (0 weeks) and post- (12 weeks) treatment visits by the 20 depression items from the Symptom Checklist 90 (Hopkins Symptom Checklist depression scale; SCL-20). Each item on the scale ranges from 0 (not at all) to 4 (extremely). Total scores are the average across all response items and range from 0 to 4 with higher scores indicating greater levels of depressive symptoms.
Time Frame: 12 Weeks
Population: One participant in the usual care group did not complete the SCL-20 at the pre-treatment visit. Therefore a change score could not be computed for this participant. The remaining number of participants in usual care for this analysis was 13.
Measure: Mean (Standard Deviation); unit: SCL-20 points
Arm/Group | Beating the Blues (BtB) | Usual Care
Number analyzed (Participants) | 7 | 13
SCL-20 points | 0.83 (0.36) | 1.44 (0.54)
Statistical Analysis 1: Comparison: Beating the Blues (BtB) vs Usual Care; Test type: Superiority; p = .019, ANCOVA; Cohen's d = 1.33

3. Secondary Outcome: Post-Treatment C-reactive Protein (CRP) Adjusted for Pre-Treatment CRP
Description: A marker of systemic inflammation measured from blood samples collected at pre- and post-treatment.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mg/l
Arm/Group | Beating the Blues (BtB) | Usual Care
Number analyzed (Participants) | 7 | 14
mg/l | 2.70 (3.15) | 4.71 (1.82)
Statistical Analysis 1: Comparison: Beating the Blues (BtB) vs Usual Care; Test type: Superiority; p = .09, ANCOVA; Cohen's d = 0.78

4. Secondary Outcome: Post-Treatment Interleukin-6 (IL-6) Adjusted for Pre-Treatment IL-6
Description: A marker of systemic inflammation measured from blood samples collected at pre- and post-treatment.
Time Frame: 12 weeks
Population: One case was excluded from the usual care group due to extreme values.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Beating the Blues (BtB) | Usual Care
Number analyzed (Participants) | 7 | 13
pg/ml | 3.76 (1.65) | 4.75 (2.84)
Statistical Analysis 1: Comparison: Beating the Blues (BtB) vs Usual Care; Test type: Superiority; p = .43, ANCOVA; Cohen's d = 0.43

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from recruitment initiation in June 2011 until study completion in July 2013. For each participant, adverse event data were collected between the pre- and post-treatment visits, for up to 12 weeks.
Arm/Group | Beating the Blues (BtB) | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/16
Other Adverse Events (participants affected / at risk) | 0/13 | 0/16

LIMITATIONS AND CAVEATS:
Missing data precluded analysis of one secondary outcome variables: Tumor Necrosis Factor-Alpha (TNF-a).

Due to the very small sample of randomized patients, conclusions should not be drawn from the results of this pilot trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes